CLINICAL TRIAL: NCT02435940
Title: Foundation Fighting Blindness My Retina Tracker Registry
Brief Title: Inherited Retinal Degenerative Disease Registry
Acronym: MRTR
Status: Recruiting | Type: Observational
Sponsor: Foundation Fighting Blindness (Other)
Responsible Party: Sponsor
Other Study IDs: FFB-Registry-01
Record Dates: First submitted 2015-04-03; First posted 2015-05-06 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Eye Diseases Hereditary; Retinal Disease; Achromatopsia; Bardet-Biedl Syndrome; Bassen-Kornzweig Syndrome; Batten Disease; Best Disease; Choroidal Dystrophy; Choroideremia; Cone Dystrophy; Cone-Rod Dystrophy; Congenital Stationary Night Blindness; Enhanced S-Cone Syndrome; Fundus Albipunctatus; Goldmann-Favre Syndrome; Gyrate Atrophy; Juvenile Macular Degeneration; Kearns-Sayre Syndrome; Leber Congenital Amaurosis; Refsum Syndrome; Retinitis Pigmentosa; Retinitis Punctata Albescens; Retinoschisis; Rod-Cone Dystrophy; Rod Dystrophy; Rod Monochromacy; Stargardt Disease; Usher Syndrome
Keywords: inherited retinal degenerative disease; retinitis pigmentosa; Usher; Leber; Bardet-Biedl; Batten; Best; cone dystrophy; cone-rod dystrophy; choroideremia; congenital night blindness; enhanced s-cone; cone monochromacy; Goldmann-Favre; Kearns-Sayre; Refsum; retinoschisis; rod-cone dystrophy; rod dystrophy; rod monochromacy; Sorsby pseudoinflammatory dystrophy; stargardt; achromatopsia; juvenile inherited macular degeneration; cone dichromacy; cone trichromacy; Charcot-Marie-Tooth; albipunctate dystrophy
MeSH Terms: conditions — Eye Diseases, Hereditary; Retinal Diseases; Color Vision Defects; Bardet-Biedl Syndrome; Abetalipoproteinemia; Neuronal Ceroid-Lipofuscinoses; Vitelliform Macular Dystrophy; Choroideremia; Cone Dystrophy; Cone-Rod Dystrophies; Night blindness, congenital stationary; Enhanced S-Cone Syndrome; Fundus Albipunctatus; Gyrate Atrophy; Stargardt Disease; Kearns-Sayre Syndrome; Leber Congenital Amaurosis; Refsum Disease; Retinitis Pigmentosa; Retinoschisis; Achromatopsia 3; Usher Syndromes; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The My Retina Tracker® Registry is sponsored by the Foundation Fighting Blindness and is for people affected by one of the rare inherited retinal degenerative diseases studied by the Foundation. It is a patient-initiated registry accessible via a secure on-line portal at www.MyRetinaTracker.org. Affected individuals who register are guided to create a profile that captures their perspective on their retinal disease and its progress; family history; genetic testing results; preventive measures; general health and interest in participation in research studies. The participants may also choose to ask their clinician to add clinical measurements and results at each clinical visit. Participants are urged to update the information regularly to create longitudinal records of their disease, from their own perspective, and their clinical progress. The overall goals of the Registry are: to better understand the diversity within the inherited retinal degenerative diseases; to understand the prevalence of the different diseases and gene variants; to assist in the establishment of genotype-phenotype relationships; to help understand the natural history of the diseases; to help accelerate research and development of clinical trials for treatments; and to provide a tool to investigators that can assist with recruitment for research studies and clinical trials.

DETAILED DESCRIPTION:
My Retina Tracker Registry provides two portals for data entry and review. Initial registration in the My Retina Tracker Registry is initiated by a participant, not a clinician. Using the participant portal, the participant establishes a username and password, is guided through on-line informed consent, and can then use an interactive guide to record their ophthalmic and family history, genotype and other subjective diagnosis-related and general health information. Drop-down menus and standardized vocabulary are used for database consistency. They may also attach documents, such as medical records, to maintain their personal medical files on their disease. Participants are encouraged to update their profiles regularly to create a longitudinal history of their disease. Participants can see aggregated data for all other participants in the registry and compare their own disease and status to others.

After a profile has been established, Registry members may ask their clinician or genetic counselor to add specific ophthalmic exam and measurement results to the profile. This is done through the clinical portal which also uses a series of drop-down menus to expedite entry and standardize data. Clinicians cannot see the participant data when adding the clinical exam data. Participants are encouraged to collect this data at each medical exam, to create a longitudinal clinical data set.

Access to de-identified data or study recruitment assistance is available to qualified investigators who may inquire by contacting Coordinator@MyRetinaTracker.org. A process that maintains patient anonymity and privacy protection, exists for researchers with Institutional Review Board-approved projects who wish to contact registry participants of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an inherited retinal degenerative disease OR

Exclusion Criteria:

* Glaucoma only
* Diabetic retinopathy only
* Non-retinal disease
* Not heritable retinal disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Affected individuals, all ages including minors registered by their parent or guardian.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2014-06; Primary Completion 2037-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Rare Diagnoses Within the Inherited Retinal Degenerative Disease Category as Defined by Clinical Evaluation | Data collection is ongoing, up to 20 years.
  Participant profiles broken out by disease category and genetic diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Todd Durham, PhD, Principal Investigator — Senior Vice President, Clinical and Outcomes Research
Locations (1):
- Foundation Fighting Blindness, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: On-line registration site for registry participants, clinicians and researchers — https://www.myretinatracker.org/
- See also: Sponsor site offers general information about rare inherited retinal degenerative diseases studied by the Foundation. — https://www.fightingblindness.org